CLINICAL TRIAL: NCT07225816
Title: Investigation of the Effect of Fasting Duration and Temporary Withholding of GLP-1 RAs on Retained Gastric Contents in Participants Treated With s.c. Liraglutide, Oral Semaglutide or s.c. Semaglutide
Brief Title: Examination of How the Duration of Fasting and Temporary Stopping of GLP-1 Medications Affect the Amount of Food Left in the Stomach in People Using Liraglutide (Injected), Semaglutide (Taken by Mouth) or Semaglutide (Injected)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9536-8438; U1111-1323-7355 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Liraglutide (Experimental): Participants will receive liraglutide subcutaneously.
  Interventions: Drug: Liraglutide
- Oral semaglutide (Experimental): Participants will receive semaglutide orally.
  Interventions: Drug: Oral Semaglutide
- Semaglutide (Experimental): Participants will receive semaglutide subcutaneously.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Liraglutide — Participants will receive liraglutide subcutaneously.
  Arms: Liraglutide
Drug: Oral Semaglutide — Participants will receive semaglutide orally.
  Arms: Oral semaglutide
Drug: Semaglutide — Participants will receive semaglutide subcutaneously.
  Arms: Semaglutide

SUMMARY:
The purpose of this study is to investigate how the duration of fasting and temporary stopping of Glucagon-Like-Peptide 1 (GLP-1) medications affect the amount of food left in the stomach in people using liraglutide (injected), semaglutide (taken by mouth) or semaglutide (injected). The length of participants participation in the study will depend on the type of GLP-1 RA treatment participants are already using.

ELIGIBILITY:
Inclusion Criteria:

- On maintenance treatment with either liraglutide 3.0 milligram (mg) for at least 5 days, oral semaglutide 25 mg for at least 5 weeks or semaglutide 2.4 mg for at least 5 weeks prior to screening.

Exclusion Criteria:

* Previous dosing in this study.
* Previous rescreening for this study.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method
* Current participation (i.e., signed informed consent) in any other interventional clinical study.
* Exposure to investigational medicinal products, except maintenance treatment with liraglutide 3.0 mg, oral semaglutide 25 mg, or semaglutide 2.4 mg as required by the inclusion criterion, within 30 days or 5 half-lives of the investigational medicinal product (if known), which-ever is longer, before screening (Visit 1).
* Any condition which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Anticipated change in lifestyle (e.g., eating, exercise or sleeping pattern) during the study.
* Participant is the investigator or other site staff or relative thereof directly involved in the conduct of the study.
* Mental incapacity, language barriers or unwillingness to comply with the requirements of the protocol, which may preclude adequate understanding or co-operation during the study as judged by the investigator.
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, or as judged by the investigator.
* History of major surgical procedures involving the oesophagus or stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) or current presence of gastrointestinal implant a*.
* Renal impairment with estimated glomerular filtration rate (eGFR) less than (<) 30 milliliter per min per 1.73 square meter (ml/min/1.73 m^2) at screening based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation according to Kidney Disease Improving Global Outcomes (KDIGO) 20246.
* Current treatment with insulin or secretagogues that might cause hypoglycaemia during periods of fasting.
* History of ketoacidosis.
* Diagnosed with or suspected to suffer from clinically significant gastroparesis, hiatal hernia or severe gastroesophageal reflux diseases with daily symptoms and/or in supine position.
* Use of other medications known to affect the motility of the stomach.
* Inability to lie in the right lateral decubitus position for gastric ultrasonography.
* Unusual meal habits and special diet requirements or unwillingness to eat the meals provided in the study.

  1. As declared by the participant or reported in the medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal after dosing of subcutaneous (s.c.) liraglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as count of participants.
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal after dosing of oral semaglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as count of participants.
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as count of participants.

SECONDARY OUTCOMES:
Gastric volume after fasting following a solid, high-fat meal after dosing of s.c. liraglutide once daily | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as milliliters per kilogram (mL/kg).
Gastric volume after fasting following a solid, high-fat meal after dosing of oral semaglutide once daily | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as mL/kg.
Gastric volume after fasting following a solid, high-fat meal after dosing of s.c. semaglutide once weekly | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as mL/kg.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal 14 days after dosing of oral semaglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as count of participants.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal after dosing of s.c. liraglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as count of participants.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 2, Day 1
  Measured as count of participants.
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal 1 day after dosing of s.c. liraglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 5
  Measured as count of participants
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal 7 days after dosing of oral semaglutide 14 mg once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 3, Day 7
  Measured as count of participants.
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal 14 days after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 14
  Measured as count of participants.
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal 2 days after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 9
  Measured as count of participants.
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal 7 days after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 5, Day 14
  Measured as count of participants.
Occurrence of empty stomach (antrum grade 0 or 1) after fasting following a solid, high-fat meal 14 days after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 6, Day 21
  Measured as count of participants.
Gastric volume after fasting following a solid, high-fat meal 1 day after dosing of s.c. liraglutide once daily | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 5
  Measured as mL/kg.
Gastric volume after fasting following a solid, high-fat meal 7 days after dosing of oral semaglutide once daily | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 3, Day 7
  Measured as mL/kg.
Gastric volume after fasting following a solid, high-fat meal 14 days after dosing of oral semaglutide once daily | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 14
  Measured as mL/kg.
Gastric volume after fasting following a solid, high-fat meal 2 days after dosing of s.c. semaglutide once weekly | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 9
  Measured as mL/kg.
Gastric volume after fasting following a solid, high-fat meal 7 days after dosing of s.c. semaglutide once weekly | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 5, Day 14
  Measured as mL/kg.
Gastric volume after fasting following a solid, high-fat meal 14 days after dosing of s.c. semaglutide once weekly | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 6, Day 21
  Measured as mL/kg.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal 1 day after dosing of s.c. liraglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 5
  Measured as count of participants.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal 7 days after dosing of oral semaglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 3, Day 7
  Measured as count of participants.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal 14 days after dosing of oral semaglutide once daily (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 14
  Measured as count of participants.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal 2 days after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 4, Day 9
  Measured as count of participants.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal 7 days after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 5, Day 14
  Measured as count of participants.
Presence of solids in the stomach (antrum grade 'solid') after fasting following a solid, high-fat meal 14 days after dosing of s.c. semaglutide once weekly (Yes/No) | 6, 8, 10, 12, 18 and 24 hours after start of fasting on Visit 6, Day 21
  Measured as count of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical LA, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: https://novonordisk-trials.com